CLINICAL TRIAL: NCT02737150
Title: CompariSon of secOnd-generation seLf-expandable Versus Balloon-expandable Valves and gEneral Versus Local Anesthesia in Transcatheter Aortic Valve Implantation (SOLVE-TAVI)
Brief Title: SecOnd-generation seLf-expandable Versus Balloon-expandable Valves and gEneral Versus Local Anesthesia in TAVI
Acronym: SOLVE-TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: University of Giessen (Other); Heart Center Leipzig - University Hospital (Other); University Hospital Schleswig-Holstein (Other); Klinikum Links der Weser Bremen (Unknown); University Hopsital Schleswig Holstein Campus Lübeck (Other); Charite University, Berlin, Germany (Other); University of Rostock (Other)
Responsible Party: Principal Investigator, Holger Thiele, MD, Director, Heart Center Leipzig - University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 15-292
Record Dates: First submitted 2016-04-05; First posted 2016-04-13 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Anesthesia, Local; Conscious Sedation; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Self-expandable valve under local anesthesia (Active Comparator): CoreValve Evolut R valve under local anesthesia with conscious sedation
  Interventions: Device: CoreValve Evolut R; Procedure: Local anesthesia with conscious sedation
- Self-expandable valve under general anesthesia (Active Comparator): CoreValve Evolut R valve under general anesthesia
  Interventions: Device: CoreValve Evolut R; Procedure: General anesthesia
- Balloon-expandable valve under local anesthesia (Active Comparator): Edwards Sapien 3 valve under local anesthesia with conscious sedation
  Interventions: Device: Edwards Sapien 3; Procedure: Local anesthesia with conscious sedation
- Balloon-expandable valve under general anesthesia (Active Comparator): Edwards Sapien 3 valve under under general anesthesia
  Interventions: Device: Edwards Sapien 3; Procedure: General anesthesia

INTERVENTIONS:
Device: CoreValve Evolut R
  Arms: Self-expandable valve under general anesthesia; Self-expandable valve under local anesthesia
Device: Edwards Sapien 3
  Arms: Balloon-expandable valve under general anesthesia; Balloon-expandable valve under local anesthesia
Procedure: Local anesthesia with conscious sedation
  Arms: Balloon-expandable valve under local anesthesia; Self-expandable valve under local anesthesia
Procedure: General anesthesia
  Arms: Balloon-expandable valve under general anesthesia; Self-expandable valve under general anesthesia

SUMMARY:
Aim of the study is to demonstrate equivalence of second-generation self-expandable valves (CoreValve Evolut R) in comparison to second-generation balloon-expandable valves (Edwards Sapien 3) and of local anesthesia with conscious sedation in comparison to general anesthesia with respect to safety and efficacy in high-risk patients with severe aortic stenosis undergoing transcatheter aortic valve implantation.

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic aortic valve stenosis defined as aortic valve area (AVA) ≤ 1cm2 or 0.6 cm²/m²
* Age ≥75 years and/or logistic European System for Cardiac Operative Risk Evaluation (EuroSCORE) ≥20% and/or Society of Thoracic Surgeons (STS) risk score ≥10% and/or high risk/contraindication to conventional surgical aortic valve replacement
* Native aortic valve annulus measuring 18-29 mm
* Suitability for transfemoral vascular access
* Written informed consent

Exclusion Criteria:

* Life expectancy <12 months due to comorbidities
* Cardiogenic shock or hemodynamic instability
* History of or active endocarditis
* Contraindications for transfemoral access
* Active peptic ulcer or upper gastro-intestinal bleeding <3 months
* Hypersensitivity or contraindication to aspirin, heparin or clopidogrel
* Contraindication for a specific mode of anesthesia as judged by the cardiac anesthesia representative of the Heart Team
* Active infection requiring antibiotic treatment
* Participation in another trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2016-04; Primary Completion 2019-02-01 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Device) | 30 day follow-up
  Number of participants with adverse events related to the treatment at 30-day follow-up consisting of all-cause mortality, stroke, moderate or severe prosthetic valve regurgitation, and permanent pacemaker implantation
Incidence of Treatment-Emergent Adverse Events (Anesthesia) | 30 day follow-up
  Number of participants with adverse events related to the treatment at 30-day follow-up consisting of all-cause mortality, stroke, myocardial infarction, infection requiring antibiotic treatment, and acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- University of Luebeck, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stachel G, Abdel-Wahab M, de Waha-Thiele S, Desch S, Feistritzer HJ, Kitamura M, Farhan S, Eitel I, Kurz T, Thiele H. Fractal dimension of the aortic annulus: a novel predictor of paravalvular leak after transcatheter aortic valve implantation. Int J Cardiovasc Imaging. 2022 Nov;38(11):2469-2478. doi: 10.1007/s10554-022-02657-1. Epub 2022 Jun 24. PMID 36434335
- [Derived] Farhan S, Stachel G, Desch S, Kurz T, Feistritzer HJ, Hartung P, Eitel I, Nef H, Doerr O, Lauten A, Landmesser U, Sandri M, Holzhey D, Borger M, Ince H, Oner A, Meyer-Saraei R, Wienbergen H, Fach A, Frey N, de Waha-Thiele S, Thiele H. Impact of moderate or severe left ventricular outflow tract calcification on clinical outcomes of patients with severe aortic stenosis undergoing transcatheter aortic valve implantation with self- and balloon-expandable valves: a post hoc analysis from the SOLVE-TAVI trial. EuroIntervention. 2022 Oct 21;18(9):759-768. doi: 10.4244/EIJ-D-22-00156. PMID 35942626
- [Derived] Feistritzer HJ, Kurz T, Stachel G, Hartung P, Lurz P, Eitel I, Marquetand C, Nef H, Doerr O, Vigelius-Rauch U, Lauten A, Landmesser U, Treskatsch S, Abdel-Wahab M, Sandri M, Holzhey D, Borger M, Ender J, Ince H, Oner A, Meyer-Saraei R, Hambrecht R, Wienbergen H, Fach A, Augenstein T, Frey N, Konig IR, Vonthein R, Funkat AK, Berggreen AE, Heringlake M, Desch S, de Waha-Thiele S, Thiele H; SOLVE-TAVI Investigators. Impact of Anesthesia Strategy and Valve Type on Clinical Outcomes After Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2021 May 4;77(17):2204-2215. doi: 10.1016/j.jacc.2021.03.007. PMID 33926657
- [Derived] Thiele H, Kurz T, Feistritzer HJ, Stachel G, Hartung P, Lurz P, Eitel I, Marquetand C, Nef H, Doerr O, Vigelius-Rauch U, Lauten A, Landmesser U, Treskatsch S, Abdel-Wahab M, Sandri M, Holzhey D, Borger M, Ender J, Ince H, Oner A, Meyer-Saraei R, Hambrecht R, Fach A, Augenstein T, Frey N, Konig IR, Vonthein R, Ruckert Y, Funkat AK, Desch S, Berggreen AE, Heringlake M, de Waha-Thiele S; SOLVE-TAVI Investigators. General Versus Local Anesthesia With Conscious Sedation in Transcatheter Aortic Valve Implantation: The Randomized SOLVE-TAVI Trial. Circulation. 2020 Oct 13;142(15):1437-1447. doi: 10.1161/CIRCULATIONAHA.120.046451. Epub 2020 Aug 21. PMID 32819145